CLINICAL TRIAL: NCT00445614
Title: Healthy, Nutritious and Tasty Fish for the Future
Brief Title: The Effects of Trout Fed With a Vegetable Based Feed on Cardiovascular Risk Markers and Plasma Proteome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Danish Institute of Fisheries Research (Other)
Responsible Party: Lotta Lauritzen, Dept. of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M187
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Disease
Keywords: nutrition; cardiovascular risk; inflammation; vascular function
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Marine trout (Experimental): 150 g/day of trout fed on marine based feed
  Interventions: Behavioral: Effects of trout on CVD risk markers and plasma proteome
- Vegetable trout (Experimental): 150 g/d of trout fed on vegetable based feed
  Interventions: Behavioral: Effects of trout on CVD risk markers and plasma proteome
- Poultry (Other): 150 g/d of poultry (for comparison)
  Interventions: Behavioral: Effects of trout on CVD risk markers and plasma proteome

INTERVENTIONS:
Behavioral: Effects of trout on CVD risk markers and plasma proteome

SUMMARY:
Fish from the aquaculture sector constitutes an increasing part of the fish consumption in Denmark. The most important farmed fish in Denmark is the rainbow trout. Due to limited access of wild fish for the feed production, alternative feeding regimes of vegetable origin such as vegetable proteins and rapeseed oil are used instead of marine feed. This change in feeding regime may affect flesh quality and health and nutritional properties as the content of long-chain n-3 polyunsaturated fatty acids (n-3 LCPUFA) will presumably decrease in the meat. The objective of the study is to investigate the effect of vegetable based feed versus marine feed of farmed trout and its effect in healthy men on cardiovascular risk markers associated with the development of cardiovascular disease (CVD).

DETAILED DESCRIPTION:
In a two month parallel study including 60 healthy men aged 40-70 years, the cardiovascular effect of one daily meal of trout fed with a vegetable based feed are compared with that of trout fed with marine feed (estimated intake of n-3 LCPUFA 2.6 g/day) and a standard Danish diet with poultry. Men are randomised to one of the three groups. Red blood cell fatty acid composition, classical cardiovascular disease (CVD)-risk markers (blood pressure and plasma lipid profile), newer CVD-markers (arterial compliance and plasma markers of endothelial function and inflammation) and plasma proteome analysis are measured at the beginning and end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Body mass index 18,5 - 30

Exclusion Criteria:

* Exercise >10 h/week
* Chronical diseases (eg. cardiovascular and diabetes)
* Regular medication
* Fish oil supplementation
* Blood donation 2 month prior or during participation
* Above maximum recommended alcohol intake
* Blood pressure >160/100 mm Hg

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
plasma protein expression
blood pressure
pulse wave analysis
pulse wave velocity
cardiovascular risk markers
markers of inflammation
plasma lipids

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, ph.d., Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrition, Denmark, Frederiksberg, Frederiksberg, Denmark